CLINICAL TRIAL: NCT07099950
Title: Dose-Dependent Functional Connectivity Effects of Low-Intensity Focused Ultrasound Applied to Deep White Matter Tracts in Humans
Brief Title: Dose-Dependent Effects of Low-Intensity Focused Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024-010
Record Dates: First submitted 2025-06-12; First posted 2025-08-01 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Healthy Controls
Keywords: Low-Intensity Focused Ultrasound; Functional Connectivity

STUDY DESIGN:
Intervention Model Description: An exploratory hypothesis is that stimulation of anteromedial structures of the telencephalic cortex of the right hemisphere and their connections with subcortical structures will lead to detectable changes in functional connectivity between these structures in a dose-dependent manner. In this study, the investigators will use a double-blind, randomized cross-over design employing either 1-LIFU or 3-LIFU. The proposed design parsimoniously follows the approved pilot study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The stimulation administration programmer will be unblinded to the type of intervention (1-epoch vs 3-epoch). Participant, study staff, and principal investigator will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dose (1-epoch) (Experimental): An 80-second train of 20-millisecond bursts of ultrasound (0.5 MHz), repeated every 200 milliseconds (400 bursts). It is estimated a 75% tissue attenuation of energy when the ultrasound wave reaches its target, therefore the investigators will set the free-field Intensity Spatial-Peak Pulse-Average (ISPPA) at 9.04 Watt /cm2 or 518 kPascal (to achieve 2.26 Watt/cm2 estimated derated ISPPA). Any modeling of actual energy delivery will be made a posteriori employing BabelBrain® software embedded in the Brainsight® neuronavigation system.
  Interventions: Other: Low-intensity focused ultrasound
- Multiple Doses (3-epoch) (Experimental): Three 80-second trains of 20-millisecond bursts of ultrasound (0.5 MHz), repeated every 200 milliseconds (400 bursts) will be administered, separated by 30 seconds each. Again, it is estimated a 75% tissue attenuation of energy when the ultrasound wave reaches its target, therefore the investigators will set the free-field Intensity Spatial-Peak Pulse-Average (ISPPA) at 9.04 Watt /cm2 or 518 kPascal (to achieve 2.26 Watt/cm2 derated ISPPA). See above for a posteriori acoustic energy modeling.
  Interventions: Other: Low-intensity focused ultrasound

INTERVENTIONS:
Other: Low-intensity focused ultrasound — 80-second stimulus with an estimated tissue ISSPA=2.26 W/cm2, administered as a single dose (1-epoch), or in multiple doses (3-epoch).

SUMMARY:
Low-intensity focused ultrasound (LIFU) has emerged as a tool to modulate the activity of deep brain structures noninvasively and reversibly, with anatomical precision. Following the results of a pilot study in which the investigators observed target engagement when LIFU was applied to the anterior limb of the internal capsule, the investigators now propose to determine the dose-response relationships of LIFU when applied to deep white matter tracts of the human brain. The investigators hope a successful study will be rapidly translatable into clinical trials seeking to understand mechanistic brain circuit-symptom relationships in major psychiatric disorders.

DETAILED DESCRIPTION:
Low intensity focused ultrasound (LIFU) is a novel technique producing noninvasive, reversible, and anatomically precise neuromodulation of deep structures in the brain. Thus far, it has been successfully employed in humans to modulate the activity of gray matter hubs, including amygdala, thalamus, and cerebral cortex. Burgeoning in vitro data shows that LIFU is also a powerful modulator of axonal conduction, by operating mechanosensitive TRAAK potassium channels in nodes of Ranvier. In a recently completed pilot study (NCT 05697172; FDA non-significant risk), the investigators translated those findings to human subjects by applying LIFU to deep brain white matter tracts, reasoning that a successful study would allow the modulation of large-scale brain circuits and thus potentially explore their mechanistic relationship with normal and abnormal behavior. Specifically, the investigators observed that a single sonication applied to tracts traversing the anterior limb of the internal capsule (ALIC) produces a functional disconnection of the connected gray matter regions, as assessed with resting state functional magnetic resonance imaging (fMRI). Now the investigators propose to define the dose-dependent effects of LIFU applied to white matter tracts regarding both intensity and duration of its neuromodulatory effects. The investigators plan to study 60 healthy adults who will be randomly exposed to two different doses of LIFU applied to tracts connecting the thalamus with the subgenual cingulate (SGCC) and orbitofrontal (OFC) cortices, namely one and three LIFU epochs (as employed in our pilot study: 80 s duration; 2.26 Watt/cm2 derated tissue peak pulse average intensity; 10% duty cycle, 500 kHz). The target white matter tracts will be defined in each individual participant by means of probabilistic tractography. The Aim 1 of this proposal is to determine the relationship between LIFU dose and intensity of target engagement in terms of decreased fMRI functional connectivity between the gray matter regions connected by the sonicated white matter tracts (i.e., thalamus and both SGCC and OFC). Aim 2 is to determine the influence of baseline structural (number of connecting streamlines) and functional (fMRI connectivity) on the dose-dependent LIFU modulation effects. In Aim 3 the investigators will determine the duration of the neuromodulation effect of the two different doses of LIFU. A successful study will result in the definition of dose-response relationships between white matter LIFU modulation and engagement of the targeted brain circuit. This will pave the way for the development of mechanistic studies consistently linking aberrant function of large-scale brain circuits and basic behavioral processes, with the long-term goal of improving the definition of precision neuromodulation targets in treatment-resistant depression and other psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* Body mass index 17-38 kg/m2.
* Fluent English speaker, capable of providing written informed consent.
* Overall Anxiety Severity and Impairment Scale <8 and Patient Health Questionnaire-9 <10
* A person of childbearing potential must have a negative urine pregnancy test at screening
* Consent that random observations of pathology are possible (e.g., brain abnormality seen during imaging).

Exclusion Criteria:

* Inability to provide informed consent including medical, psychiatric, or other conditions that restrict the patient's following abilities: to interpret the study information, to give informed consent, to adhere to the rules of the protocol, or complete the study.
* No telephone or easy access to telephone
* Has active suicidal ideation (as measured by Suicide-Risk-Assessment-C-SSRS "Yes" answers to items 3, 4, or 5 Suicidal Ideation-Past 1 month section, or any "Yes" answer to any of the items of Suicidal Behavior-Past 3 months section), or any suicide attempt in the last 3 months
* Has positive test result(s) for alcohol of abuse (including methadone, opiates, cocaine, amphetamine/methamphetamine and ecstasy), or substance use disorder including alcohol, stimulants, sedatives, and cannabis exceeding mild severity in the last 6 months
* Has a lifetime APA Diagnostic and Statistical Manual of Mental Disorders (DSM)-5th edition including major depression, generalized anxiety disorder, specific phobias, panic disorder, post-traumatic stress disorder, schizophrenia spectrum and other psychotic disorders, obsessive-compulsive disorder, or bipolar disorder.
* Benzodiazepines or anticonvulsants in the 7 days prior to participation.
* MRI contradictions as detected by the MRI Safety Screen including claustrophobia and unwillingness and inability to complete scans (e.g., unable to lie on one's back for 60 mins.
* Clinical history of relevant structural pathology of the central nervous system, including Parkinson's disease, multiple sclerosis, and brain malignant neoplasia.
* History of unstable liver or renal insufficiency; significant and unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, hematological, rheumatological, or metabolic disturbance; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit or confound the protocol-specified assessments, including uncontrolled diabetes mellitus (ss evidenced by fasting glycemia ≥ 120 mg/dL or hemoglobin A1c ≥ 6.5%) or hypertension (as evidenced by two consecutive readings ≥ 140/90 mmHg) to ensure medical stability throughout this longitudinal study.
* Moderate-to-severe traumatic brain injury or any other clinical neurocognitive disorder.
* Clinical history of at least minor neurocognitive disorder of any origin.
* Prescription of a medication outside of the accepted range, as determined by best clinical practices and current research.
* Use of any psychotropic medication.
* Unwillingness or inability to complete any major aspects of the study protocol.
* Prior neurosurgery.
* Non-correctable vision or hearing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post-Sonication Changes in Tissue Engagement | Pre- vs up to 30 minutes post-sonication for 1-epoch vs 3-epoch LIFU.
  Changes in resting-state functional (fMRI) connectivity (FC) between thalamus and both subgenual (sgCC) and orbitofrontal (OFC) cortices after one vs. after three-epoch LIFU.

SECONDARY OUTCOMES:
Post-Sonication Changes in Functional Connectivity with Respect to Structural Connectivity | Pre- vs up to 30 minutes post-sonication for 1-epoch vs 3-epoch LIFU.
  Establishment of a Pearson correlation between the number of thalamo-OFC and thalamo-sgCC streamlines, and resting-state fMRI FC changes between the thalamus and OFC or sgCC regions, respectively, after one- and three-LIFU epoch stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No